CLINICAL TRIAL: NCT03912701
Title: If Early Warning Systems Were Used, Could the Risk of Early Clinical Deterioration be Predicted and Re-admission to Intensive Care Could be Prevented
Brief Title: Early Warning Systems, Risk of Early Clinical Deterioration
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Erzincan University (Other)
Responsible Party: Principal Investigator, ILKE KUPELI, assist. prof., Erzincan University
Other Study IDs: EBYU 3
Record Dates: First submitted 2019-04-09; First posted 2019-04-11 (Actual); Last update posted 2019-07-17 (Actual); Status verified 2019-07

CONDITIONS: Early Clinical Deterioration
MeSH Terms: conditions — Clinical Deterioration

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Vitalpac early warning score (VIEWS) — The Vitalpac early warning score (ViEWS) is an early warning system aimed primarily at prediction of the first 24-hour mortality in emergency patients and has not been used to assess intensive care unit discharge.

SUMMARY:
Primary purpose of the study was to evaluate the relationship between "NEWS" and "VIEWS" scores of patients who were screened retrospectively, early clinical deterioration, return to intensive care and morbidity / mortality.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years
* patients who were taken back to the intensive care unit in the first 24 hours

Exclusion Criteria:

* under 18 years old,
* patients undergoing postoperative intensive care,
* pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over the age of 18 and discharged and admitted to intensive care in the first 24 hours
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-08-01 (Estimated); Primary Completion 2019-11-01 (Estimated); Study Completion 2019-11-15 (Estimated)

PRIMARY OUTCOMES:
Number of patients who were taken back to intensive care unit due to early clinical deterioration | six month
  Number of patients who were taken back to intensive care unit due to early clinical deterioration

CONTACTS AND LOCATIONS:
Locations (1):
- Erzincan University, Erzincan, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kaben A, Correa F, Reinhart K, Settmacher U, Gummert J, Kalff R, Sakr Y. Readmission to a surgical intensive care unit: incidence, outcome and risk factors. Crit Care. 2008;12(5):R123. doi: 10.1186/cc7023. Epub 2008 Oct 6. PMID 18838006
- [Result] Prytherch DR, Smith GB, Schmidt PE, Featherstone PI. ViEWS--Towards a national early warning score for detecting adult inpatient deterioration. Resuscitation. 2010 Aug;81(8):932-7. doi: 10.1016/j.resuscitation.2010.04.014. PMID 20637974
- [Result] McGinley A, Pearse RM. A national early warning score for acutely ill patients. BMJ. 2012 Aug 8;345:e5310. doi: 10.1136/bmj.e5310. No abstract available. PMID 22875955